CLINICAL TRIAL: NCT04972201
Title: The Performance of a Pan-cancer Early Detection Model Based on Liquid Biopsy of Various-omics Biomarkers: a Proof of Concept Study
Brief Title: A Proof of Concept Study of Pan-cancer Early Detection by Liquid Biopsy
Acronym: PROMISE
Status: Completed | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Guangzhou Burning Rock Dx Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: RSCD2020006
Record Dates: First submitted 2021-07-15; First posted 2021-07-22 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2021-06

CONDITIONS: Cancer
Keywords: cancer; liquid biopsy; cell-free DNA (cfDNA); microRNA (miRNA); early detection
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer Arm: Participants with new diagnosis of cancer, from whom blood samples will be collected.
  Interventions: Device: Multi-cancer early detection test
- Healthy Arm: Participants without known presence of malignancies or benign diseases, from whom blood samples will be collected.
  Interventions: Device: Multi-cancer early detection test

INTERVENTIONS:
Device: Multi-cancer early detection test — Blood collection and multi-cancer early detection test

SUMMARY:
PROMISE is a multi-center, prospective and proof of concept study aimed to evaluate the performance of 3 prototype assays of cell-free DNA (cfDNA) mutation, cfDNA methylation and microRNA (miRNA) expression in early detection of multi-cancer. Assay(s) will be selected for further development. The study will enroll approximately 2035 participants, including participants with cancers and healthy participants.

DETAILED DESCRIPTION:
Blood samples will be prospectively collected from cancer patients and non-cancer individuals. Targeted cell-free DNA (cfDNA) methylation panel of ~490,000 CpG sites, a 168-gene mutation panel and 16 proteins will be applied. Participants will be stratified by age and clinical status and split into the training and the testing sets. The multi-cancer detection blood test models were developed on training set and validated on testing set.

ELIGIBILITY:
Inclusion Criteria for Cancer Arm Participants:

* Ability to provide a written informed consent
* 40-75 years old
* Ability to comply with study procedures
* Confirmed diagnosis or suspicious cases of one of the 9 types of cancers within 42 days prior to study blood draw.
* No prior anti-cancer therapy (local or systematic) prior to study blood draw

Exclusion Criteria for Cancer Arm Participants:

* Pregnancy or lactating women
* Recipients of organ transplant or prior non-autologous (allogeneic) bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 7 days prior to study blood draw
* Recipients of any anti-cancer therapy within 30 days prior to study blood draw, due to diseases other than cancer
* Known prior diagnosis of malignancies, other current malignant diseases or multiple primary tumors
* No confirmed diagnosis of cancer by histopathological or radiological assessments within 42 days of study blood draw, or diagnosis of a benign disease or precancerous lesions by histopathological assessments, or inability to characterize whether the lesion is malignant or benign

Inclusion Criteria for Healthy Arm Participants:

* Ability to provide a written informed consent
* 40-75 years old
* No cancer-related symptoms or discomfort within 30 days prior to study blood draw
* Ability to comply with study procedures
* No clinically significant finding by laboratory tests and radiology examinations

Exclusion Criteria for Healthy Arm Participants:

* Pregnancy or lactating women
* Recipients of organ transplant or prior non-autologous (allogeneic) bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 7 days prior to study blood draw
* Clinically significant or uncontrolled comorbidities
* Prior or ongoing treatment of cancer within 3 years prior to study blood draw

Ages: 40 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be re recruited from medical centers and assigned into two arms, including participants with new diagnosis of cancers and healthy participants.
Sampling Method: Non-Probability Sample
Enrollment: 2305 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity of early detection of cancers and Tissue of origin (TOO) accuracy of 3 assays of cfDNA mutation, cfDNA methylation and miRNA expression when specificity was 90%, 95% or 98% in healthy participants | 9 months
  Sensitivity of early detection of cancers and Tissue of origin (TOO) accuracy of 3 assays of cfDNA mutation, cfDNA methylation and miRNA expression when specificity was 90%, 95% or 98% in healthy participants

SECONDARY OUTCOMES:
Sensitivity, specificity and TOO accuracy of an assay of cfDNA mutation in various types of cancer in different stages | 9 months
  Sensitivity, specificity and TOO accuracy of an assay of cfDNA mutation in various types of cancer in different stages
Sensitivity, specificity and TOO accuracy of an assay of cfDNA methylation in various types of cancer in different stages | 9 months
  Sensitivity, specificity and TOO accuracy of an assay of cfDNA methylation in various types of cancer in different stages
Sensitivity, specificity and TOO accuracy of an assay of miRNA expression in various types of cancer in different stages | 9 months
  Sensitivity, specificity and TOO accuracy of an assay of miRNA expression in various types of cancer in different stages
Sensitivity, specificity and TOO accuracy of combined assays of cfDNA mutation, cfDNA methylation and/or miRNA expression in early detection of cancers | 9 months
  Sensitivity, specificity and TOO accuracy of combined assays of cfDNA mutation, cfDNA methylation and/or miRNA expression in early detection of cancers

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, M.D., Ph.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No